CLINICAL TRIAL: NCT06342752
Title: The Role of Volatile Organic Compounds (VOCs), Airway Mucins and Microbiome in the Development of Bronchopulmonary Dysplasia and the Feasibility of Exhaled Breath VOCs Analysis as an Early Detection Tool
Brief Title: The Role of Volatile Organic Compounds (VOCs), Airway Mucins and the Microbiome in the Early Prediction of Bronchopulmonary Dysplasia (BPD)
Acronym: INFANCY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: 6007
Record Dates: First submitted 2024-03-13; First posted 2024-04-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Volatile Organic Compounds; Preterm birth; Airway microbiome; Airway mucins; Exhaled breath analysis; Placental microbiome; Vaginal microbiome; Early prediction of BPD; Inflammation Lungs; Respiratory morbidity; multiple breath washout test
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Pneumonia | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preterm infants: all included infants will undergo a breath test and two throat swabs, in case the infant is intubated also endotracheal aspirates will be collected
  Interventions: Diagnostic Test: Breath test; Other: Throat swabs; Other: Endotracheal aspirates
- Mothers of preterm infants: placental biopsies, a placental swab and a vaginal swab will be taken after birth
  Interventions: Other: Placental samples; Other: Vaginal swab

INTERVENTIONS:
Diagnostic Test: Breath test — Early detection of volatile organic compounds (VOCs) in breath from preterm infants, collected at several timepoints within the first 4 weeks of life to predict BPD before diagnosis is made at 36 weeks PMA.
  Other Names: Exhaled breath analysis; Volatomics; Exhaled Volatile Organic Compounds; Exhaled VOCs
  Groups: Preterm infants
Other: Throat swabs — A throat swab will be taken on several timepoints within the first 4 weeks of life to detect airway mucin expression. A second throat swab will be taken as proxy for the airway microbiome.
  Groups: Preterm infants
Other: Placental samples — After birth, placental biopsies will be collected for headspace VOCs analysis. A placental swab and a biopsy will be taken for microbiome analysis.
  Other Names: Placental headspace VOCs analysis; Placental swabs
  Groups: Mothers of preterm infants
Other: Vaginal swab — A vaginal swab will be taken before birth for microbiome analysis.
  Groups: Mothers of preterm infants
Other: Endotracheal aspirates — Collection of aspirates, as part of routine care, to detect mucin expression and the lung microbiome.
  Other Names: Aspirates
  Groups: Preterm infants

SUMMARY:
Bronchopulmonary dysplasia (BPD), the most common respiratory complication of extremely preterm birth, significantly impacts healthcare with high morbidity and mortality rates.

Despite the well-established primordial role of inflammation and oxidative stress in the development of BPD, clinical practice does not incorporate the testing for biomarkers associated with the development of BPD. The diagnosis of BPD based on required respiratory support at 36 weeks PML, stresses the need for an early prediction tool which could identify patients with high levels of these biomarkers. This on its turn, could also improve treatment approaches in clinical practice which are currently mostly supportive or non-specific and do not target underlying pathophysiologic pathways.

Secondly, mucin expression aim to play a rol in other respiratory diseases, whereas in BPD only the potential role of MUC1 was explored.

Thirdly, the composition of the airway microbial composition of an infant is assumed to be influenced by different factors. From early on in pregnancy the airway microbiome of the infant is formed, offering a protective role against pathologies. On the other hand, the role of the airway microbiome in the development of BPD remains unclear and needs to be elucidated.

The threefold aim of this study is as follows:

I. The development of a non-invasive breath test that allows early detection of bronchopulmonary dysplasia, using the potential of VOCs in exhaled breath as biomarkers for inflammation and oxidative stress.

II. The exploration of the composition and diversity of the airway microbiome in infants with BPD, their association with exhaled VOCs and the exploration of the placental and vaginal microbiome.

III. The detection of potential alterations in airway mucin expression in BPD patients.

Through this comprehensive approach, we seek to gain a deeper understanding of how these mutual associations may contribute to the later development of BPD.

In total 140 preterm infants, including 70 BPD patients and 70 preterm controls, born below 30 weeks' gestation at the Antwerp University Hospital will be included.

DETAILED DESCRIPTION:
After birth, a swab and samples will be collected from the placenta, next to a maternal vaginal swab for microbiome analysis. Breath samples, two oropharyngeal swabs and endotracheal aspirates - in case intubated - will be collected from the infant on different days in the first 28 days of life.

At 36 weeks PMA, BPD is diagnosed if the infant still requires respiratory support. An oxygen reduction test will also be performed to determine if the infant can maintain saturations within a predetermined target range (90-96% in our hospital) during a stepwise reduction of oxygen, while closely monitoring the neonate. At 36 weeks PMA, infants diagnosed with BPD - as well as controls - will undergo a one-time capillary (or venous) blood gas test, which will be mostly done as part of routine care. The blood gas test will be combined with a continuous transcutaneous capnography (tcPCO2) for 24 hours to assess the degree of severity of lung damage, i.e. grade of alveolar hypoventilation by means of hypercapnia.

All enrolled participants, regardless of BPD diagnosis, will have two clinical follow-up study visits after discharge to home, at 6 and at 12 months corrected age. Another oropharyngeal swab will be collected at these visits for microbiome analysis. To assess lung function in all BPD patients, a multiple breath washout test during natural sleep after the administration of melatonin, will be performed at 6 and 12 months corrected age. At 6 and 12 months corrected age, a chest CT will be performed in severe BPD-cases to assess lung structure. Results of follow-up investigations, clinical data, as well as respiratory questionnaires will be used to correlate to findings of the analysis of all samples taken in the NICU. With this approach, it is not only possible to explore if possible biomarkers found in the early weeks of life could predict BPD at 36 weeks PML, but also respiratory/pulmonary outcome at 6 and 12 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* Born at a gestational age < 30 weeks

Exclusion Criteria:

* Major congenital defect or disorder
* Patients with an unstable general condition as deemed by the attending neonatologist

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborn infants born preterm < 30 weeks gestational age at the Antwerp University Hospital and admitted to the neonatal intensive care unit.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Exhaled breath Volatile Organic Compounds (VOCs) | first 4 weeks of life
  Abbundance of VOCs in breath samples to distinguish BPD from preterm controls by means of GC-MS: direct samples in the respiratory circuit as well as indirect samples from air in the incubator
Vaginal microbiome | right before delivery
  Metagenomic shotgun sequencing after extraction of bacterial DNA from vaginal swabs after birth
Placental microbiome | at delivery
  Metagenomic shotgun sequencing after extraction of bacterial DNA from samples and subamniotic swabs after birth
Placental headspace VOCs | at delivery
  Abbundance of VOCs in the headspace of placental samples to distinguish BPD from preterm controls
Airway mucin profiles | first 4 weeks of life
  Genetic expression of airway mucins in BPD and preterm controls on oropharyngeal samples via qRT-PCR
Airway microbial profiles | 12 months
  16S RNA sequencing or metagenomic shotgun sequencing after extraction of bacterial DNA from oropharyngeal swabs and aspirates in BPD and preterm controls

SECONDARY OUTCOMES:
Hypercapnia | 3 months
  BPD patients will undergo a blood gas test to assess the degree of lung damage severity
Follow-up structural lung imaging | 12 months
  Chest CT scan in severe BPD cases
Pulmonary function | 12 months
  To determine lung function - as an objective outcome parameter - a multiple breath washout (MBW) test will be performed, all infants with BPD, at the corrected age of 6 and 12 months.
Chronic lung disease outcome 6 months corrected age | 6 months
  Validated respiratory questionnaire will be completed by the parents at 6 months corrected age. The questionnaire at 6 months is based on the Liverpool Respiratory Symptom Questionnaire (LRSQ), a validated tool for evaluating the prevalence of common paediatric respiratory symptoms amongst preschool children. It consists of eight domains, each containing between three and five items. The first six domains assess respiratory symptoms and the remaining two assess the impact of symptoms on the child and family.
Chronic lung disease outcome 12 months corrected age | 12 months
  At 12 months the validated questionnaire 'A parent-completed respiratory questionnaire for 1-year-old children' will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Antonius Mulder, MD, PhD,prof, Principal Investigator — University Hospital Antwerp, Belgium; Stijn L Verhulst, MD, PhD,prof, Study Director — University Hospital Antwerp, Belgium
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No